CLINICAL TRIAL: NCT06944080
Title: Effect of Deep Margin Elevation With Different Base Materials on Fracture Resistance of Direct and Indirect Resin Composite Restorations and Periodontal Health(Clinical and Experimental Studies)
Brief Title: Effect of Different Base Materials on Ginigiva During Gingival Margin Elevation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Rofida Ragab Mohamed, Assistant lecturer in operative department, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: gingival marginal elevation
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-01

CONDITIONS: Gingival Margin Elevation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The effect of deep Margin elevation with different base materials on periodontal health (Experimental): The effect of deep Margin elevation with different base materials (resin modified glass ionomer, flowable composite, injectable hybrid composite) on periodontal health (in vivo study)will be applied then plaque index, gingival index, probing depth, clinical attachment level and biochemical marker will be measured at base line and after 3 months
  Interventions: Other: base material(Tetric® N-Flow,Beautifil-Flow PLUS,GC fuji II LC capsule)

INTERVENTIONS:
Other: base material(Tetric® N-Flow,Beautifil-Flow PLUS,GC fuji II LC capsule) — subgingival restoration, deep marginal elevation procedure with different base materials will be applied then plaque index, gingival index, probing depth, clinical attachment level and biochemical marker will be measured at base line and after 3 months.

SUMMARY:
This study will be conducted to investigate

1. The effect of deep margin elevation with different base materials (resin modified glass ionomer, flowable composite, injectable hybrid composite) on fracture resistance and marginal quality of direct and indirect resin composite inlay (in vitro).
2. The effect of deep margin elevation with different base materials (resin modified glass ionomer, flowable composite, injectable hybrid composite) on periodontal health (in vivo study).

DETAILED DESCRIPTION:
The dental clinician has consistently challenged the restoration of deep proximal lesions since they are usually associated with significant defects with subgingival margins exceeding cementoenamel junction (CEJ).

In this clinical scenario, indirect restorations are preferable since they provide better esthetic, anatomic form, physical and mechanical properties, and reduced polymerization shrinkage due to their extraoral fabrication that permits the relief of residual stresses .

However, subgingival margins remain a challenge as they are challenging to handle due to limited access, rubber dam slippage over the margin, and subsequent persistent saliva, crevice fluid and blood leakage.

The conventional approach includes orthodontic extrusion, surgical exposure of the cervical margin, or a combination of both techniques leading to an apical displacement of supporting tissues to access the subgingival margin and obtain adequate space for the establishment of biological width (BW).

Frequently, these techniques mentioned above may cause further attachment loss and exposure of root concavities and furcation's to the oral environment, dentin hypersensitivity, and unfavorable crown to root ratio as well as compromised esthetics. Additionally, this process may often delay the delivery of the final restoration.

An alternative and more conservative approach, the so-called "deep margin elevation" (DME), is to apply a base over the preexisting cervical margin to relocate it coronally.

This technique introduced in 1998 by Dietschi and Spreafico is also referred to with the terms "cervical margin relocation", "proximal box elevation", and "coronal margin relocation", and presents several benefits concerning proper isolation with a rubber dam and subsequent moisture control, facilitation in impression taking, proper bonding procedures, and excess removal and avoidance of unnecessary tissue sacrifice.

The open-sandwich technique is widely considered the forerunner of DME introduced to overcome sealing issues in deep Class II direct composite restorations, the open-sandwich technique uses a glass ionomer or resin-modified glass ionomer (RM-GIC) to fill the cervical part of the box, which results in a part of the glass ionomer/resin-modified glass ionomer being exposed to the oral environment.

However, even if the two techniques resemble each other, DME was initially described for indirect restorations using composite resin. The adhesive composite resin base is used to seal the dentin, correct geometry, reinforce undermined cusps, and fill undercuts.

Flowable composite bases and liners may also act as stress absorbers or stress breakers during the insertion and polymerization of subsequent layers or during functional loading. Beside other physical properties, the elastic modulus of the restorative material plays a major role for the stress-absorbing effect.

RM-GIC releases fluoride, hydrophilic nature, flexibility, chemical bonding and enhanced mechanical and wear properties of their newer generations, could be a more suitable option for bonding to deep moist dentin/cementum margins.

A base, liner, and final restorative all in one; Beautifil Flow Plus is the next step in the evolution of restorative materials, combining the convenience of a flowable delivery system with strength and functionality that surpass leading hybrid composites, superior adaptation ensures a tight marginal seal, decreasing voids, high radiopacity allows clear visibility during follow-ups and Fluoride release and recharge is ideal for high caries index patients.

When the marginal ridges are involved in large lesions; it is wise to plan for indirect restorations (IRs), the strength of the tooth is directly proportional to the integrity of the marginal ridges. Depending on the extent of tooth structure loss, the need for cuspal coverage and the amount of reinforcement needed.

IRs such as inlays, onlays, overlays and full-contour crowns are recommended. Historically, IRs fabricated using gold alloys were considered the gold standard. However, due to increased demand for more natural and esthetic restorations, the use of composites and ceramics have overhauled the use of metals.

Fracture is considered the most common reason for replacing fixed partial prostheses. For this reason, when considering the long-term viability of a dental material for fabricating restorations, it is essential to test its fracture resistance.

So, this study will be conducted to investigate the effect of proximal box elevation at different depth level with three base materials (resin modified glass ionomer, flowable composite and injectable hybrid composite) and its influence on fracture resistance of premolars teeth restored with direct and indirect composite inlay.

The null hypothesis tested that there is no significant difference in the effect of deep margin elevation with (RM-GI and Flowable composite) base materials on fracture resistance and marginal quality of direct and indirect resin composite when compared to injectable hybrid composite.

ELIGIBILITY:
Inclusion Criteria:

* good oral hygien
* upper premolar teeth

Exclusion Criteria:

* badly destructed tooth

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The effect of deep Margin elevation with different base materials (resin modified glass ionomer, flowable composite, injectable hybrid composite) on periodontal health (in vivo study) | base line
  after subgingival restoration(resin modified glass ionomer, flowable composite, injectable hybrid composite) will be applied to to elevate deep marginal then biochemical marker will be measured (TNF,IL-1 by pg/ml) from gingival crevicular fluid.

SECONDARY OUTCOMES:
The effect of deep Margin elevation with different base materials (resin modified glass ionomer, flowable composite, injectable hybrid composite) on periodontal health (in vivo study) | after 3 months
  follow up after 3 months of subgingival restoration(resin modified glass ionomer, flowable composite, injectable hybrid composite) will be applied to to elevate deep marginal to measure level of biochemical marker in gingival crevicular fluid (TNF,IL-1 by pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: ahmed abdallah khalil, Study Director — Faculty of dentistry-Minia university; rasha saad zaghlool, Study Director — Faculty of dentistry-Minia university